CLINICAL TRIAL: NCT01681901
Title: Lymph Node Evaluation in the Axilla of Symptomatic Older Women During Breast Sonography.
Brief Title: Ultrasound in Detecting Lymph Node Metastasis in Older Patients Undergoing Breast Sonography
Status: Withdrawn | Type: Observational
Why Stopped: no patient accrual
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: OSU-06010; NCI-2012-01176 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-09-05; First posted 2012-09-10 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Diagnostic (ultrasound): Patients undergo breast ultrasound imaging.
  Interventions: Procedure: ultrasound imaging

INTERVENTIONS:
Procedure: ultrasound imaging — Undergo ultrasound
  Other Names: ultrasonography; ultrasound; ultrasound test

SUMMARY:
This pilot clinical trial studies ultrasound in detecting lymph node metastasis in older patients with undergoing breast sonography. Diagnostic procedures, such as ultrasound, may help find breast cancer and find out how far the disease has spread

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To develop a reliable and consistent set of guidelines for utilizing diagnostic ultrasound to assess axillary lymph nodes for patient suspicious of breast cancer with possible nodal metastasis.

SECONDARY OBJECTIVES:

I. To explore whether the data collected can be used for pathologic validation of metastatic disease.

OUTLINE:

Patients undergo breast ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for a breast ultrasound
* Patients who have had a mammogram with a Breast Imaging Reporting and Data System (BIRADS) of >= 4
* Patients who are undiagnosed for breast cancer

Exclusion Criteria:

* Patients who have had breast cancer surgery

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion Criteria:
  * Patients referred for a breast ultrasound
  * Patients who have had a mammogram with a Breast Imaging Reporting and Data System (BIRADS) of >= 4
  * Patients who are undiagnosed for breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-06-07 (Actual); Primary Completion 2007-04 (Estimated); Study Completion 2007-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of successful evaluations, defined as the consistent capture of the data for geometry, morphology, qualitative vascular information, and quantitative vascular information on 3 axillary lymph nodes | at 15 minutes following breast sonogram
  The proposed methodology will be considered unfeasible if the proportion of successful evaluations is =< 0.7.

SECONDARY OUTCOMES:
Accuracy of lymph node geometry, measured with a longitudinal and transverse ratio, to determine guidelines for characterizing micro metastases to the lymph nodes | 3 months
  Descriptive statistics, such as means, proportions and standard deviations, will be summarized. The longitudinal-transverse ratio will be investigated for cutoff points that yield high sensitivity and to see if results are consistent with prior studies suggesting a ratio of 1.5 or less is indicative of abnormality. The percent agreement between the resulting diagnostic criteria and the surgical/pathological results will be assessed.
Accuracy of lymph node morphology, assessed for shape and echogenicity, to determine guidelines for characterizing micro metastases to the lymph nodes | 3 months
  Descriptive statistics, such as means, proportions and standard deviations, will be summarized. The percent agreement between the resulting diagnostic criteria and the surgical/pathological results will be assessed.
Accuracy of lymph node vascularity, assessed with color doppler, to determine guidelines for characterizing micro metastases to the lymph nodes | 3 months
  Descriptive statistics, such as means, proportions and standard deviations, will be summarized. The percent agreement between the resulting diagnostic criteria and the surgical/pathological results will be assessed.
Accuracy of lymphatic flow, measured with spectral doppler, to determine guidelines for characterizing micro metastases to the lymph nodes | 3 months
  Descriptive statistics, such as means, proportions and standard deviations, will be summarized. The percent agreement between the resulting diagnostic criteria and the surgical/pathological results will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Evans, Principal Investigator — Ohio State University Comprehensive Cancer Center

REFERENCES:
- See also: The Jamelsine — http://cancer.osu.edu